CLINICAL TRIAL: NCT02036580
Title: A Phase 2, Multicenter, Double-Blind Within Cohort, Dose-escalation Study to Evaluate the Safety and Tolerability of Multiple Doses of CAT-354 (Tralokinumab) in Japanese Patients With Idiopathic Pulmonary Fibrosis
Brief Title: D2212C00002 J-Phase II Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D2212C00002
Record Dates: First submitted 2014-01-13; First posted 2014-01-15 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-01

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Japan; Phase2; Safety; Tolerability; Idiopathic Pulmonary Fibrosis; IPF; CAT-354; Tralokinumab
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Low Dose (Experimental): Investigational product Tralokinumab
  Interventions: Biological: tralokinumab cohort 1
- High Dose (Experimental): Investigational product Tralokinumab
  Interventions: Biological: tralokinumab cohort 2
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: tralokinumab cohort 1 — Tralokinumab is a human recombinant monoclonal antibody (MAb) of the subclass that specifically binds human IL-13, blocking interactions with the IL-13 receptor
  Arms: Low Dose
Biological: tralokinumab cohort 2 — Tralokinumab is a human recombinant monoclonal antibody (MAb) of the subclass that specifically binds human IL-13, blocking interactions with the IL-13 receptor
  Arms: High Dose
Other: Placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of multiple-doses of tralokinumab in Japanese patients with Idiopathic Pulmonary Fibrosis.

DETAILED DESCRIPTION:
This is a phase II, multicenter, blinded within cohort, dose-escalation study to evaluate the safety and tolerability of two ascending doses of tralokinumab in Japanese patients aged ≥ 50 years with mild to moderate Idiopathic Pulmonary Fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* Confirmed IPF diagnosis for ≤ 5 years prior to Visit 1 (screening). Confirmation of diagnosis of IPF
* Mild to moderate IPF to include all of the following at Visit 1

  1. FVC ≥ 50% and ≤ 90% predicted normal
  2. Partial pressure of oxygen in arterial blood (PaO2) of ≥ 55 mmHg on room air, or oxygen saturation by pulse oximetry (SpO2) of ≥ 90% on room air at rest
  3. Hemoglobin-corrected diffusion capacity for carbon monoxide (DLCO) ≥ 30% and ≤ 90% predicted normal

Exclusion Criteria:

* History of clinically significant environmental exposure (eg, domestic and occupational) to a known cause of pulmonary fibrosis
* Diagnosis of connective tissue disease or drug toxicity as the likely cause of the interstitial disease
* A suspected IPF exacerbation not fully resolved and treatment completed ≤ 14 days prior to Visit 1
* A suspected IPF exacerbation during the screening period
* A FEV1/FVC ratio < 0.70 at the time of Visit 1 (postbronchodilator)
* The extent of emphysema on the HRCT is greater than the extent of fibrosis

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph M Parker, MD, Study Director — MedImmune LLC
Locations (5):
- Japan (5):
  - Research Site, Fukuoka
  - Research Site, Himeji-shi
  - Research Site, Seto-shi
  - Research Site, Shibuya-ku
  - Research Site, Yokohama

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 37 patients were screened at 5 centres in Japan, and 20 patients were randomized and received at least 1 dose of tralokinumab low dose, high dose, or placebo.
  The first patient entered the study on 24 January 2014 and the last patient last visit was on 19 November 2015.
Pre-assignment Details: 20 patients were randomized and received at least 1 dose of tralokinumab low dose, high dose, or placebo (tralokinumab low dose group: n=8, tralokinumab high dose group: n=8, placebo group: n=4).
Groups:
- Low Dose: Tralokinumab 400 mg Q4W intravenously dosed for 24 weeks
- High Dose: Tralokinumab 800 mg Q4W intravenously dosed for 24 weeks
- Placebo: Placebo Q4W intravenously dosed for 24 weeks
Period: Overall Study
Arm/Group | Low Dose | High Dose | Placebo
Started | 8 | 8 | 4
Completed | 7 | 7 | 4
Not Completed | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose | High Dose | Placebo | Total
Number analyzed (Participants) | 8 | 8 | 4 | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.0 (7.1) | 65.0 (9.4) | 68.3 (8.5) | 66.5 (8.0)
Gender [Count of Participants; unit: Participants]
  Female | 2 | 2 | 0 | 4
  Male | 6 | 6 | 4 | 16

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability Primarily Assessed by the Number of Patients With Adverse Events
Description: Adverse events and serious adverse events using the Safety Population. Other variables used for the safety assessments include electrocardiogram, vital signs, and routine laboratory assessments. These variables as well as their changes from baseline will be summarized descriptively.
Time Frame: From baseline to Week 48 (treatment-emergent only)
Population: Safety population
Measure: Number; unit: Patients
Arm/Group | Low Dose | High Dose | Placebo
Number analyzed (Participants) | 8 | 8 | 4
Patients
  At lease one adverse events | 8 | 7 | 2
  At least one IP related adverse event | 1 | 2 | 0
  At least one adverse event of ≥ grade 3 severity | 1 | 0 | 0
  Death (grade 5 severity) | 0 | 0 | 0
  At least one serious adverse event | 2 | 1 | 1
  At least one serious and ≥ grade 3 severity event | 0 | 0 | 0
  At least one IP related serious adverse event | 0 | 0 | 0
  At least one event leading to IP discontinuation | 2 | 0 | 0

2. Secondary Outcome: Serum Tralokinumab Concentration Data
Description: Serum tralokinumab concentration data will be summarized by treatment group.
Time Frame: From baseline to Week 48 (Week 0 [post-dose, within +5 minutes after end of infusion], Week 4 [pre-dose], Week 12 [pre-dose]. Week 28, Week 40, Week 48)
Population: PK population
Measure: Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | Low Dose | High Dose
Number analyzed (Participants) | 8 | 8
Microgram per milliliter
  Week 0 (post-dose) | 149 (64.8) | 313 (46.6)
  Week 4 (pre-dose) | 33.9 (9.03) | 76.1 (32.3)
  Week 12 (pre-dose) | 55.1 (16.1) | 75.7 (41.8)
  Week 28 | 61.4 (29.1) | 87.5 (50.9)
  Week 40 | 2.55 (2.70) | 2.69 (1.72)
  Week 48 | 0.515 (0.759) | 0.374 (0.270)

3. Secondary Outcome: Immunogenecity
Description: The incidence rate of positive serum antibodies to tralokinumab will be reported.
Time Frame: From baseline to Week 48
Population: Safety population
Measure: Number; unit: Patients
Arm/Group | Low Dose | High Dose | Placebo
Number analyzed (Participants) | 8 | 8 | 4
Patients
  Anti-drug antibody positive at baseline | 1 | 0 | 0
  Anti-drug antibody positive post-baseline | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From baseline to Week 48 (treatment-emergent only)
Arm/Group | Low Dose | High Dose | Placebo
Serious Adverse Events (participants affected / at risk) | 2/8 | 1/8 | 1/4
Other Adverse Events (participants affected / at risk) | 8/8 | 7/8 | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose (N=8) | High Dose (N=8) | Placebo (N=4)
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose (N=8) | High Dose (N=8) | Placebo (N=4)
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Chronic gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | 0
Noninfective gingivitis (Gastrointestinal disorders) | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 2 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 4 | 1 | 1
Pharyngitis (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 1
Blood pressure increased (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Formication (Nervous system disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 2 | 0
Calculus ureteric (Renal and urinary disorders) | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Intermittent claudication (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No